# **DET VIDENSKABSETISKE KOMITÉSYSTEM**

#### Det Videnskabsetisk Komitésystem

**(S3)** 

#### Informed consent for participating in a clinical trial

Research project title:

A combined treatment with GM-CSF, fosfomycin and metronidazole for pouchitis in ulcerative colitis patients after restorative ileal pouch anal anastomosis surgery

A clinical safety and proof-of-concept study .

Participant information version 4 - English Phase 1

En kombinationbehandling med GM-CSF, fosfomycin og metronidazol mod pouchitis ved colitisulcerosa patienter, efter ileal-pouch analanstomose. Et klinisk sikkerheds- og pilotstudie

Phase 1 study

Trial narticinant's name.

### Statement from the trial participant:

I have received written and verbal information and I know and understand enough about the reason, methods, benefits and disadvantages of this trial to agree to participate.

I know that it is voluntary to participate in this trial, and that I at any point in time can retract my consent without losing my current and future rights to treatment.

I give consent to participate in this clinical trial, and that biological material is taken for storage in a research biobank. I have received a copy of this informed consent form as well as a copy of written information about this project for my own use.

| That participant 5 name. |
|---|
| Date:Signature |
| Would you like to be informed about the trial's results as well as whether this has any consequences for you? |
| Yes(put an x) No(put an x) |
| Statement from the one that gives trial information: |
| I declare that the trial participant has received verbal and written information about the trial. |
| In my belief there has been given sufficient information so that the participant can decide whether ornot to participate in the clinical trial. |
| Name of the person giving information: Viviane Lin, MD |
| Date:Signature: |
| EudraCT nr: 2020-000609-10 |

Informed Consent version 1

### **(S3)**

#### Informed consent for participating in a clinical trial

Research project title:

A combined treatment with GM-CSF, fosfomycin and metronidazole for pouchitis in ulcerative colitis patients after restorative ileal pouch anal anastomosis surgery

A clinical safety and proof-of-concept study .

En kombinationbehandling med GM-CSF, fosfomycin og metronidazol mod pouchitis ved colitis ulcerosa patienter, efter ileal-pouch analanstomose. Et klinisk sikkerheds- og pilotstudie

Phase 2 study

## Statement from the trial participant:

Trial participant's name:

I have received written and verbal information and I know and understand enough about the reason, methods, benefits and disadvantages of this trial to agree to participate.

I know that it is voluntary to participate in this trial, and that I at any point in time can retract my consent without losing my current and future rights to treatment.

I give consent to participate in this clinical trial, and that biological material is taken for storage in a research biobank. I have received a copy of this informed consent form as well as a copy of written information about this project for my own use.

| · · · | |
|---|---|
| Date: | Signature |
| Would you like to be info you? | rmed about the trial's results as well as whether this has any consequences for |
| Yes(put an x) No_ | (put an x) |
| Statement from the one that gives trial information: | |
| I declare that the trial par | ticipant has received verbal and written information about the trial. |
| In my belief there has been given sufficient information so that the participant can decide whether or not to participate in the clinical trial. | |
| Name of the person giving information: Viviane Lin, MD | |
| Date:S | ignature: |

EudraCT nr: 2020-000609-10

Participant Information Version 4 – English Phase 2